CLINICAL TRIAL: NCT06223893
Title: CirrhoCare, A Real-world, Randomised Controlled Study, to Determine the Clinical and Cost-effectiveness of CirrhoCare Digital Home Monitoring and Management in Patients With Decompensated Cirrhosis
Brief Title: CirrhoCare- Using Smart-phone Technology to Enhance Care and Access to Treatment for Cirrhosis
Acronym: CirrhoCare
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: CyberLiver Ltd (Unknown); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 151197
Record Dates: First submitted 2023-10-31; First posted 2024-01-25 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Decompensated Cirrhosis

STUDY DESIGN:
Intervention Model Description: Participants will be randomised 1:1 to receive either the standard of care or the CirrhoCare management system.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CirrhoCare management system (Other)
  Interventions: Device: CirrhoCare management system
- Standard of Care (No Intervention)

INTERVENTIONS:
Device: CirrhoCare management system — This is a UKCA-marked, digital-therapeutic system consisting of:
  * clinical-grade, cirrhosis monitoring sensors and a smartphone app,
  * a clinical team-facing, decision-facilitating dashboard, and
  * CyberLiver's platform incorporating hepatic algorithms.
  The CirrhoCare kit consists of: - Apple watch - iPhone with an in-built CirrhoCare app - a digital Bluetooth-linked system comprised of: ~Wellue BP monitor, ~Wellue weighing scale ~Bluetooth thermometer.
  The CirrhoCare management system also includes:
  * The clinician dashboard: All participant data collected through the app will be reviewed by the clinical team via the clinician dashboard.
  * The CirrhoCare algorithm: This algorithm will advise the clinical team if the participant is at high, medium, or low risk of developing a particular outcome event, based on monitoring data collected each day from the participant which is compared to the baseline values and average values collected over the first week of monitoring.
  Arms: CirrhoCare management system

SUMMARY:
The CirrhoCare trial is a multi-centre, open label randomised controlled trial in patients with decompensated cirrhosis. The trial aims to investigate the clinical and cost-effectiveness of CirrhoCare digital home monitoring and management with current standard of care in these patients.

DETAILED DESCRIPTION:
Cirrhosis, progressive scaring of the liver- has many causes, principally, excessive alcohol intake, fatty-liver and viral infections. Unlike many chronic diseases, cirrhosis deaths are increasing rapidly year-on-year. It is the third commonest cause of premature, UK working-age deaths, with 62,000 years of working-life lost each year and NHS care costs of £4.53bn annually. One quarter of all UK cirrhosis patients are at-risk of acute decompensation, whereby complications such as fluid-overload, confusion and infections arise, requiring hospital-emergency treatment.

Currently, decompensated cirrhosis patients require regular hospital clinical assessments to detect these new complications. Even following hospital discharge, readmission with new decompensating complications approaches 37% in 4 weeks. This disease burden, compounded by increasing alcohol and obesity-driven liver disease, means demand for specialist liver services outweighs current capacity in a resource-stretched healthcare system. Moreover, regional variation of specialist liver services also impacts on illness and deaths, leading to a postcode lottery of care access and geographical inequity.

The CirrhoCare trial, addresses this urgent clinical-need through an innovative cirrhosis management system, including home-monitoring of decompensated cirrhosis patients, measuring vital signs such as heart rate and blood pressure (using low cost, sensing technology), assessing weight (smart-scale) and mental ability (smartphone app), all of which are impacted as cirrhosis progresses. By efficiently and securely collecting data on CyberLiver's management-system (platform), CirrhoCare provides a decision-facilitating tool, incorporating individual-patient data, helping liver-physicians to optimise and personalise treatment in the community.

The CirrhoCare trial investigators also plan to assess clinical and cost effectiveness of CirrhoCare management and seek regulatory approvals. This innovative aspect of cirrhosis management will be more acceptable and convenient for patients. It will also deliver community care with environmental, sustainable benefits, through reduced hospital visits, despite increasing service demands. The cost- effectiveness analysis will generate value-for-money evidence of CirrhoCare management, and the clinical evidence needed to inform future adoption into the NHS.

ELIGIBILITY:
Inclusion criteria:

1. Adults ≥ 18 years and diagnosed with cirrhosis of any aetiology.
2. Cirrhosis defined by standard clinical criteria, ultrasonographic findings and/or histology. Cirrhosis of any aetiology may be included. However, participants with cirrhosis due to autoimmune hepatitis must be on a stable corticosteroid dose for ≥3-month period before study inclusion (to be recorded on concomitant log).
3. Cirrhosis severity-risk defined by European-Foundation Consortium Liver Failure - Acute Decompensation score (CLIF-C AD score) ≥42 points but ≤65 points at the time of screening.
4. Hospitalisation for acute decompensation [determined as one or more of the following: increasing ascites, variceal haemorrhage, overt hepatic encephalopathy, spontaneous bacterial peritonitis (SBP) or hepatorenal syndrome - acute kidney injury (HRS-AKI)].
5. Participants able to give informed consent.

Exclusion criteria:

1. Participants with ACLF grade 2 and above according to the criteria published by Moreau
2. Participants with CLIF-C AD score ≥ 66, who have a high mortality similar to ACLF ≥2 participants.
3. Current overt hepatic encephalopathy, defined as grade II-IV hepatic encephalopathy according to the West-Haven classification, unable to give consent.
4. Participants with active hepatocellular carcinoma (HCC) or history of HCC that is in remission for less than six months for uninodular HCC or for less than 12 months for multinodular HCC within Milan criteria.
5. Participants with a history of significant extra hepatic disease with impaired short-term prognosis, including congestive heart failure New York Heart Association Grade III/IV, COPD GOLD >2, chronic kidney disease with serum creatinine >2mg/dL or under renal replacement therapy.
6. Participants with documented refractory ascites on a palliative pathway.
7. Participants who are active on the transplant waiting list.
8. Participants with current extra hepatic malignancies including solid tumours and hematologic disorders.
9. Participants with mental incapacity, significant language barriers, or any other reason considered by the investigator precluding adequate understanding, cooperation or compliance in the study.
10. Participants with active viral infections, or yet to achieve clear response to anti-viral therapy.
11. Any disorders likely to impact on study engagement, including severe frailty, severe addiction history (including opioids) with evidence of multiple recent relapses.
12. Any other reason that the PI considers would make the participant unsuitable to enter CirrhoCare (e.g., participants on an end-of-life palliative care pathway).
13. Participants enrolled in other interventional trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2023-11-24 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Number of hospital interventions from new-liver related complications | 90 days from randomisation
  The CirrhoCare trial will investigate whether the CirrhoCare management system leads to a reduction in the requirement for unplanned medical intervention from new-liver related complications over 90 days from hospital discharge.

SECONDARY OUTCOMES:
Effects on CLIF-C AD score | 90 days from randomisation
  To determine the effects of the CirrhoCare management system on the Chronic Liver Failure Consortium Acute Decompensation (CLIF-C AD) score. [Minimum score is 0 and there is no upper limit. The higher the score the worse the outcome)
Effects on MELD score | 90 days from randomisation
  To determine the effects of the CirrhoCare management system on the Model for End-Stage Liver Disease score ( MELD). [Score ranges from 6-40. The higher the score the worse the outcome]
To determine the effects of the CirrhoCare management system on the number of liver-related deaths at 90 days | 90 days from randomisation
  To determine the effects of the CirrhoCare management system on the number of liver-related deaths at 90 days.
Healthcare resource use analysis | 90 days from randomisation
  To assess healthcare resource use through analysis of the number of healthcare appointments during the study period
Healthcare cost analysis | 90 days from randomisation
  To assess the financial costs associated with healthcare interventions during the study period (measured in British Pound Sterling).
User experience and engagement | 90 days from randomisation
  To assess user experience and engagement through questionnaires and interviews : The questionnaires will be graded from 1-10 for each question, with 0 is extremely negative as a response, and 10 very highly positive response.
Quality of Life (EQ-5D-5L) assessment | 90 days from randomisation
  To assess health-related quality of Life through the EuroQol 5-Dimension 5-Level (EQ-5D-5L) questionnaire. The score ranges from -0.59 to 1, with a score of 1 representing the best possible health status.
Frailty assessment | 90 days from randomisation
  To assess frailty using the Liver Frailty Index. The score ranges from 1.0 to 7.0 with higher scores representing increased levels of frailty.
Mortality | 90 days from randomisation
  To assess mortality (overall survival)
Number of hospital readmissions | 90 days from randomisation
  To assess the overall number of readmissions to hospital
Effects of the individual components making up the primary outcome | 90 days from randomisation
  Assessment of the effects of the individual components making up the primary outcome. Each complication of cirrhosis will be individually assessed between CirrhoCare and standard of care groups. [Ascites based on Gr 1-3 and HE based on West Haven criteria 1-4; Infection Positive or Negative culture]
Longitudinal effects of all secondary outcomes | Day 28, Day 56, Day 90
  The longitudinal effects of all secondary outcomes will be investigated by using an appropriate model that incorporates the Day 28 and Day 56 visits in addition to the Day 90 visit
Length of hospital readmissions | 90 days from randomisation
  Assessment of the length of stay for each hospital readmission for a given participant recorded in days.

OTHER OUTCOMES:
Nutritional impact analysis | 90 days from randomisation
  To assess whether there is a change in nutritional status using the Royal Free Hospital Nutrition Prioritizing Tool (RFH-NPT). The score ranges from 0-7, with higher scores being associated with an increased risk of malnutrition.

CONTACTS AND LOCATIONS:
Overall Officials: Rajeshwar Mookerjee, Study Chair — UCL
Locations (15):
- United Kingdom (15):
  - The Royal London Hospital, Barts Health NHS Trust, London, London
  - Queen Elizabeth Hospital Birmingham, University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Royal Sussex County Hospital, University Hospitals Sussex NHS Foundation Trust, Brighton
  - Walsgrave General Hospital, University Hospital Coventry & Warwickshire NHS Trust, Coventry
  - Royal Liverpool University Hospital, Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - Whittington Hospital, Whittington Health NHS Trust, London
  - Royal Free Hospital, Royal Free London NHS Foundation Trust, London
  - St Thomas Hospital, Liverpool University Hospitals NHS Foundation Trust, London
  - King's College Hospital, King's College Hospital NHS Foundation Trust, London
  - St George's Hospital, St George's university Hospital NHS Foundation Trust, London
  - Queen's Medical Centre, Nottingham University Hospitals NHS Trust, Nottingham
  - John Radcliff Hospital, Oxford University Hospitals NHS Foundation Trust, Oxford
  - Derriford Hospital, University Hospitals Plymouth NHS Trust, Plymouth
  - Southampton General Hospital, University Hospital Southampton NHS Foundation Trust, Southampton
  - Torbay Hospital, Torbay and South Devon NHS Foundation Trust, Torquay